CLINICAL TRIAL: NCT03823885
Title: E-Cigarettes and Monocytes
Brief Title: ECigs, Inflammation and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Principal Investigator, Holly R Middlekauff, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 18001147
Record Dates: First submitted 2019-01-24; First posted 2019-01-31 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: E-cigarettes, Oxidative Stress, Inflammation
MeSH Terms: conditions — Vaping; Inflammation | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Crossover with 2 week washout
Who Masked: Outcomes Assessor
Masking Description: Code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-cig (Experimental): One time exposure to e-cig
  Interventions: Other: e-cigarette
- sham (Experimental): One time exposure to empty e-cig
  Interventions: Other: empty (-cigarette sham control)

INTERVENTIONS:
Other: e-cigarette — use e-cig for 30 minutes
  Other Names: e-cig
  Arms: E-cig
Other: empty (-cigarette sham control) — use empty e-cig (sham control)
  Other Names: empty e-cig
  Arms: sham

SUMMARY:
Randomized controlled trial of acute use of electronic cigarette effect on oxidative stress and inflammation.

DETAILED DESCRIPTION:
Participants will have an acute e-cig exposure on 2 occasions 1) e-cigarette 2) sham e-cig (empty e-cig) control. Blood will be collected before and after E-cig use and analyzed for biomarkers of inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Cardiac disease Respiratory disease Diabetes

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Cellular Reactive Oxygen Species, units = % fluorescence | within 4 hours of E-cig use
  cellular oxidative stress, including cytoplasmic and mitochondrial oxidative stress, in viable cells

SECONDARY OUTCOMES:
CD 14+ Monocyte, units = % of total cells | within 4 hours of e-cig use
  CD 14+ Monocyte, % of total cells will be measured with antibodies and stable dye

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kelesidis T, Tran E, Arastoo S, Lakhani K, Heymans R, Gornbein J, Middlekauff HR. Elevated Cellular Oxidative Stress in Circulating Immune Cells in Otherwise Healthy Young People Who Use Electronic Cigarettes in a Cross-Sectional Single-Center Study: Implications for Future Cardiovascular Risk. J Am Heart Assoc. 2020 Sep 15;9(18):e016983. doi: 10.1161/JAHA.120.016983. Epub 2020 Sep 8. PMID 32896211